CLINICAL TRIAL: NCT04553042
Title: A Single-Dose, Open-Label, Randomized, Crossover Study to Assess the Bioequivalence Between Different Formulations and Phase 3 Formulation of Seltorexant Under Fasted Conditions in Healthy Participants
Brief Title: A Study of Seltorexant in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CR108883; 42847922MDD1018 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-09-14; First posted 2020-09-17 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — seltorexant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment Sequence ABC (Experimental): Participants will receive a single dose of seltorexant as formulation (Test 1) (Treatment A) in Treatment Period 1, followed by a single dose of seltorexant as formulation (Test 2) (Treatment B) in Treatment Period 2, followed by a single dose of seltorexant as formulation (Reference) (Treatment C) in Treatment Period 3 on Day 1 of each Treatment Period under fasted condition. There will be a washout period of 7 to 14 days from dosing on Day 1 of each Treatment Period.
  Interventions: Drug: Seltorexant
- Treatment Sequence BCA (Experimental): Participants will receive Treatment B in Treatment Period 1, followed by Treatment C in Treatment Period 2, followed by Treatment A in Treatment Period 3 on Day 1 of each Treatment Period under fasted condition. There will be a washout period of 7 to 14 days from dosing on Day 1 of each Treatment Period.
  Interventions: Drug: Seltorexant
- Treatment Sequence CAB (Experimental): Participants will receive Treatment C in Treatment Period 1, followed by Treatment A in Treatment Period 2, followed by Treatment B in Treatment Period 3 on Day 1 of each Treatment Period under fasted condition. There will be a washout period of 7 to 14 days from dosing on Day 1 of each Treatment Period.
  Interventions: Drug: Seltorexant
- Treatment Sequence CBA (Experimental): Participants will receive Treatment C in Treatment Period 1, followed by Treatment B in Treatment Period 2, followed by Treatment A in Treatment Period 3 on Day 1 of each Treatment Period under fasted condition. There will be a washout period of 7 to 14 days from dosing on Day 1 of each Treatment Period.
  Interventions: Drug: Seltorexant
- Treatment Sequence ACB (Experimental): Participants will receive Treatment A in Treatment Period 1, followed by Treatment C in Treatment Period 2, followed by Treatment B in Treatment Period 3 on Day 1 of each Treatment Period under fasted condition. There will be a washout period of 7 to 14 days from dosing on Day 1 of each Treatment Period.
  Interventions: Drug: Seltorexant
- Treatment Sequence BAC (Experimental): Participants will receive Treatment B in Treatment Period 1, followed by Treatment A in Treatment Period 2, followed by Treatment C in Treatment Period 3 on Day 1 of each Treatment Period under fasted condition. There will be a washout period of 7 to 14 days from dosing on Day 1 of each Treatment Period.
  Interventions: Drug: Seltorexant

INTERVENTIONS:
Drug: Seltorexant — Seltorexant will be administered orally as per assigned treatment sequence.
  Other Names: JNJ-42847922

SUMMARY:
The purpose of this study is to evaluate the bioequivalence of Test 1 and/or Test 2 seltorexant tablet formulations with respect to Reference seltorexant tablet formulation in healthy participants receiving a single dose under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Be healthy on the basis of medical history (screening only), physical examination, vital signs, and 12-lead electrocardiogram (ECG) performed at screening and Day-1 of Treatment Period 1 or prior to randomization
* Be healthy on the basis of clinical laboratory tests performed at screening
* All female participants (regardless of childbearing potential), must have a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test at screening and a negative urine pregnancy test on Day-1 of each treatment period
* Body mass index (BMI) between 18.0 and 30.0 kilogram per meter square (kg/m^2, inclusive (BMI = weight/height^2), and body weight not less than 50 kilogram (kg)
* Blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeter of Mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency (estimated glomerular filtration rate [eGFR] less than (<) 80 milliliter per minute (mL/min)/1.73 per meter square (m^2) at screening only), thyroid disease, neurologic (including seizure disorders) or psychiatric disease (depression or anxiety disorder in remission and no longer requiring medication is acceptable), infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results. Significant past gastrointestinal medical history, or any disease/surgery that would with interfere drug absorption
* Has any significant or is suspected to have a primary sleep disorder, including but not limited to obstructive sleep apnea, restless leg syndrome, or parasomnias based on history and/or physical exam. Participants with insomnia disorder are allowed if not requiring medication
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for acetaminophen, oral contraceptives, and hormonal replacement therapy within 14 days before the first dose of the study drug is scheduled
* Known allergies, hypersensitivity, or intolerance to seltorexant or its excipients
* Positive test for human immunodeficiency virus (HIV)-1 and HIV-2 antibodies, hepatitis B surface antigen (HbsAg), or hepatitis C antibodies at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Seltorexant and its Metabolites | Predose, up to 48 hours post dose (Day 3)
  Cmax is defined as the maximum observed plasma concentration of seltorexant and its metabolites.
Last Observed Measurable Plasma Concentration (Clast) of Seltorexant and its Metabolites | Predose, up to 48 hours post dose (Day 3)
  Clast is defined as the last observed measurable (non-below quantification limit [non-BQL]) plasma concentration of seltorexant and its metabolites.
Time to Reach the Maximum Observed Plasma Concentration (Tmax) of Seltorexant and its Metabolites | Predose, up to 48 hours post dose (Day 3)
  Tmax is defined as the actual sampling time to reach the maximum observed plasma concentration of seltorexant and its metabolites.
Area Under the Concentration-time Curve From Time Zero to Time of the Last Measurable Plasma Concentration (AUC [0-last]) of Seltorexant and its Metabolites | Predose, up to 48 hours post dose (Day 3)
  AUC (0-last) is defined as area under the plasma concentration-time curve from the time of dosing to the last measurable plasma concentration of seltorexant and its metabolites.
Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUC [0-infinity]) of Seltorexant and its Metabolites | Predose, up to 48 hours post dose (Day 3)
  AUC (0-infinity) is defined as area under the plasma concentration-time curve of seltorexant and its metabolites extrapolated to infinity, calculated using the linear trapezoidal method from time zero to infinite time calculated as the sum of AUC(0-last)+C(last)/ lambda(z).
Apparent Terminal Elimination Half-life (t1/2) of Seltorexant and its Metabolites | Predose, up to 48 hours post dose (Day 3)
  Apparent elimination half-life associated with the terminal slope lambda(z) of the semilogarithmic drug concentration-time curve of seltorexant and its metabolites.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) including AEs of Special Interest (AESI) as a Measure of Safety and Tolerability | Up to 11 Weeks
  Number of participants with an AE including AE of special interest as a measure of safety and tolerability will be reported. An AE is any untoward medical occurrence in a clinical study participant administered a investigational or non-investigational medicinal product. An AE does not necessarily have a causal relationship with the treatment. AESI will comprise of cataplexy, sleep paralysis, complex, sleep-related behaviors/parasomnias, sleep terrors, bruxism, sleep sex, sleep related eating disorder, sleep behavior disorder, catathrenia and abnormal (vivid) dreams.
Number of Participants with Laboratory Abnormalities | Up to 11 Weeks
  Number of participants with laboratory abnormalities related to hematology, serum chemistry, coagulation, and urinalysis will be reported.
Number of Participants with Clinically Significant Changes in Vital Signs | Up to 11 Weeks
  Number of participants with clinically significant changes in vital signs including blood pressure, heart rate, respiratory rate, oral temperature will be reported.
Number of Participants with Abnormalities in Electrocardiogram (ECG) | Up to 11 Weeks
  Number of participants with abnormalities in ECG will be reported.
Number of Participants with Clinically Significant Changes in Physical Examination | Up to 11 Weeks
  Number of participants with clinically significant changes in physical examination including height and body weight will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA Health Sciences, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency